CLINICAL TRIAL: NCT07294846
Title: Drug Interaction Study on Linaprazan Glurate Capsules, Clarithromycin Tablets, Amoxicillin Capsules, and Bismuth Potassium Citrate Capsules
Brief Title: Drug Interaction Study on Linaprazan Glurate Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Sinorda Biomedicine Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SND-X842-103
Record Dates: First submitted 2025-09-04; First posted 2025-12-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers; Patients
Keywords: Potassium competitive acid blocker; Acid inhibition; Adjunctive therapy for H. pylori eradication; PK; Linaprazan Glurate Capsules
MeSH Terms: interventions — Amoxicillin; Clarithromycin; Esomeprazole

STUDY DESIGN:
Intervention Model Description: This study investigates the drug-drug interactions (DDI) among Linaprazan Glurate capsules, clarithromycin tablets, amoxicillin capsules, and bismuth potassium citrate capsules. The research plan is divided into two parts: a study in Hp-negative healthy subjects and a study in Hp-positive subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Linaprazan Glurate Capsules 50mg BID, consecutive 7-day dosing per period (Experimental): Glurate Capsules Capsules 50mg, BID, consecutive 7-day dosing per period in Part 1.
  Interventions: Drug: Linaprazan Glurate Capsules; Drug: Amoxicillin Capsules; Drug: Clarithromycin tablets
- Linaprazan Glurate Capsules 50mg BID, consecutive 14-day dosing (Experimental): Linaprazan Glurate Capsules 50mg BID, consecutive 14-day dosing in part 2.
  Interventions: Drug: Linaprazan Glurate Capsules; Drug: Bismuth Potassium Citrate Capsules; Drug: Amoxicillin Capsules; Drug: Clarithromycin tablets
- Esomeprazole Magnesium Enteric-coated Tablets 20mg BID, consecutive 14-day dosing. (Experimental): Esomeprazole Magnesium Enteric-coated Tablets 20mg, BID in Part 2.
  Interventions: Drug: Bismuth Potassium Citrate Capsules; Drug: Amoxicillin Capsules; Drug: Clarithromycin tablets; Drug: Esomeprazole Magnesium Enteric-coated Tablets

INTERVENTIONS:
Drug: Linaprazan Glurate Capsules — Linaprazan Glurate capsules
  Other Names: Linaprazan Glurate
  Arms: Linaprazan Glurate Capsules 50mg BID, consecutive 14-day dosing; Linaprazan Glurate Capsules 50mg BID, consecutive 7-day dosing per period
Drug: Bismuth Potassium Citrate Capsules — Bismuth Potassium Citrate Capsules
  Other Names: Bismuth Potassium Citrate
  Arms: Esomeprazole Magnesium Enteric-coated Tablets 20mg BID, consecutive 14-day dosing.; Linaprazan Glurate Capsules 50mg BID, consecutive 14-day dosing
Drug: Amoxicillin Capsules — Amoxicillin Capsules
  Other Names: Amoxicillin
Drug: Clarithromycin tablets — Clarithromycin Tablets
  Other Names: Clarithromycin
Drug: Esomeprazole Magnesium Enteric-coated Tablets — Esomeprazole Magnesium Enteric-coated Tablets
  Other Names: Esomeprazole Magnesium
  Arms: Esomeprazole Magnesium Enteric-coated Tablets 20mg BID, consecutive 14-day dosing.

SUMMARY:
This study is a drug-drug interaction (DDI) investigation involving Linaprazan Glurate capsules and a combination of clarithromycin tablets, amoxicillin capsules, and bismuth potassium citrate capsules. The study plan is divided into two parts: one involving Hp-negative healthy subjects and the other involving Hp-positive subjects.

DETAILED DESCRIPTION:
The first part of the study is designed as a single-center, randomized, open-label, four-period, four-sequence crossover trial to evaluate the changes in pharmacokinetic (PK) profiles of Linaprazan Glurate capsules when co-administered with clarithromycin tablets and amoxicillin capsules compared to their individual administration, as well as the safety and tolerability of the combination therapy in Hp-negative healthy adult Chinese subjects.

The second part of the study is designed as a single-center, randomized, open-label, parallel-group, positive-controlled trial to compare the differences in systemic exposure of bismuth potassium citrate capsules between the Linaprazan Glurate capsule-based quadruple therapy (combined with clarithromycin tablets, amoxicillin capsules, and bismuth potassium citrate capsules) and the esomeprazole magnesium enteric-coated tablet-based quadruple therapy (combined with clarithromycin tablets, amoxicillin capsules, and bismuth potassium citrate capsules), to evaluate the pharmacodynamic effects on intragastric pH, to assess the safety and tolerability of the Linaprazan Glurate capsule-based quadruple therapy, and to preliminarily explore its efficacy in eradicating Helicobacter pylori (Hp) in Hp-positive subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18 to 55 years old (including 18 and 55);
2. Male weight ≥50.0 kg, female weight ≥45.0 kg; Body Mass Index (BMI) between 19.0 and 26.0 kg/m²(including critical value); BMI=weight/height2 (m2)
3. Part 1 Study and Part 2 Study:

   Part 1: Subjects must be Helicobacter pylori-negative at screening; Part 2: Subjects must be Helicobacter pylori-positive at screening;
4. From signing informed consent until 3 months after study completion, subjects must: Implement appropriate and effective contraception to prevent pregnancy (applies to subject or partner); Refrain from sperm donation or egg donation plans;
5. Subjects must fully comprehend the trial content, voluntarily participate in the trial, Provide written informed consent;

Exclusion Criteria:

1. Subjects known as Hypersensitivity History: Known allergy to: Linaprazan Glurate capsules, Esomeprazole (Part 2 only), Penicillin, Macrolide antibiotics, Any component of bismuth potassium citrate;History of severe immediate hypersensitivity to: Other macrolide antibiotics, β-lactam agents (e.g., cephalosporins, carbapenems, monobactams),Multiple drug hypersensitivity (e.g., allergic reactions to ≥2 medications/foods);
2. Clinically Significant Abnormalities at Screening: Abnormalities deemed clinically significant by investigators based on: Medical history review, Vital signs, Physical examination, 12-lead ECG, Laboratory tests: Complete blood count (CBC), Blood chemistry, Urinalysis, Coagulation tests ;
3. Subjects with Penicillin sodium skin test positivity during screening;
4. Subjects with use of any investigational product within 3 months prior to screening;
5. Subjects with use of potassium-competitive acid blockers (P-CABs) within 3 months prior to screening;
6. Subjects with use within 30 days prior to screening of Prescription drugs, Over-the-counter ,OTC) medications, Herbal medicines, Dietary supplements;
7. Subjects with history of diseases in the following systems (also investigator-determined as ineligible): Central nervous system, Cardiovascular system, Respiratory system, Digestive system, Endocrine system, Immune system, Neurological/Psychiatric systems, Hematologic/Lymphatic systems, Musculoskeletal system;
8. Gastrointestinal/Surgical History: History of gastrointestinal diseases or surgeries including:Gastric surgery (except pyloromyotomy for infantile pyloric stenosis), Cholecystectomy, Vagotomy, Bowel resection, Any surgery potentially affecting GI motility, pH, or absorption, Conditions impacting drug ADME: Dysphagia, Vomiting, Severe diarrhea;
9. Cardiac Abnormalities: Clinically significant ECG abnormality history, Family history of Long QT Syndrome (grandparents, parents, siblings), Screening QTcF prolongation: 450 msec in males, 470 msec in females;
10. Subjects with major surgery within 3 months prior to screening,and planned surgery during trial participation;
11. Subjects with blood donation (whole blood/component) ≥400 mL within 3 months (excluding menstrual loss),Blood transfusion or blood product use within 3 months;
12. Infectious Disease Screening: Positive results for any at screening: Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCV-Ab), HIV antibody (HIV-Ab), Treponema pallidum antibody (TP-Ab);
13. Subjects who have used illicit drugs within the 3 months prior to screening, or have a history of drug abuse within the past 12 months, or whose urine drug abuse screening test result is positive;
14. Subjects who regularly consumed alcohol within the 3 months prior to screening (i.e., consuming more than 14 standard units per week; 1 unit = 360mL of beer, or 45mL of 40% spirits, or 150mL of wine), or who are unwilling to abstain from alcohol or any alcohol-containing products for 48 hours prior to dosing and during the trial, or whose alcohol breath test result is positive;
15. Subjects who smoked an average of >5 cigarettes per day within the 30 days prior to screening; or who cannot guarantee abstinence from smoking from the signing of the informed consent form until the end of the study;
16. Subjects who have been vaccinated within the 3 months prior to screening or plan to be vaccinated during the trial period;
17. Subjects who consumed excessive amounts of tea, coffee, or caffeinated beverages (more than 8 cups per day; 1 cup = 250mL) within the 4 weeks prior to screening;
18. Subjects who consumed special diets (including pitaya, mango, grapefruit, pomelo, lime, starfruit, or foods/beverages prepared from them, or any caffeinated foods/beverages, alcoholic beverages, or other foods/beverages known to affect drug absorption, distribution, metabolism, or excretion) within 48 hours prior to the first dose;
19. Subjects who are intolerant to venipuncture, have difficulty with blood collection, or have a history of needle or blood phobia/syncope;
20. Pregnant or lactating women;
21. Subjects with special dietary requirements who cannot comply with the standardized diet, or who have difficulty swallowing;
22. Subjects deemed unsuitable for participation by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2025-09-08 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Steady state maximum concentration (Cmax,ss) | 7 days
  Cmax,ss of of Linaprazan Glurate and its active metabolite(s), clarithromycin and its active metabolite(s), and amoxicillin in Part 1 study.
AUC0-τ,ss(The area under the drug-time curve within the dosing interval after reaching the steady state) | 7 days
  AUC0-τ,ss of Linaprazan Glurate and its active metabolite(s), clarithromycin and its active metabolite(s), and amoxicillin in Part 1 study.
Cav,ss (Average steady-state blood drug concentration) | 7 days
  Cav,ss of Linaprazan Glurate and its active metabolite(s), clarithromycin and its active metabolite(s), and amoxicillin in Part 1 study.
Tmax,ss (Steady-state peak time) | 7 days
  Tmax,ss of Linaprazan Glurate and its active metabolite(s), clarithromycin and its active metabolite(s), and amoxicillin in Part 1 study.
CLss/F(Steady-state apparent clearance rate) | 7 days
  CLss/F of Linaprazan Glurate and its active metabolite(s), clarithromycin and its active metabolite(s), and amoxicillin in Part 1 study.
t1/2z(Terminal elimination half-life) | 7, 14 days
  t1/2z of Linaprazan Glurate and its active metabolite(s), clarithromycin and its active metabolite(s), and amoxicillin in Part 1 study; and t1/2z of Pharmacokinetic Parameters of Bismuth in Part 2 study.
Vz/F (Apparent volume of distribution in the terminal elimination phase) | 7, 14 days
  Vz/F of Linaprazan Glurate and its active metabolite(s), clarithromycin and its active metabolite(s), and amoxicillin in Part 1 study; and Vz/F of Pharmacokinetic Parameters of Bismuth in Part 2 study.
λz (Terminal elimination rate constant) | 7, 14 days
  λz of Linaprazan Glurate and its active metabolite(s), clarithromycin and its active metabolite(s), and amoxicillin in Part 1 study; and λz of Pharmacokinetic Parameters of Bismuth in Part 2 study.
MRT(mean residence time) | 7 days
  MRT of Linaprazan Glurate and its active metabolite(s), clarithromycin and its active metabolite(s), and amoxicillin in Part 1 study.
Cmax(Maximum observed plasma drug concentration) | 14 days
  Cmax of Pharmacokinetic Parameters of Bismuth in Part 2 study.
AUC0-τ (The area under the drug-time curve within the dosing interval) | 14 days
  AUC0-τ of Pharmacokinetic Parameters of Bismuth in Part 2 study.
Tmax (Time to reach maximum plasma concentration) | 14 days
  Tmax of Pharmacokinetic Parameters of Bismuth in Part 2 study.
CL/F (apparent clearance) | 14 days
  CL/F of Pharmacokinetic Parameters of Bismuth in Part 2 study.
Ae0-τ (Amount of drug excreted in urine over the dosing interval) | 14 days
  Ae0-τ of Pharmacokinetic Parameters of Bismuth in Part 2 study.
fe (Amount of drug excreted in urine over the dosing interval) | 14 days
  fe of Pharmacokinetic Parameters of Bismuth in Part 2 study.
CLR (renal clearance) | 14 days
  CLR of Pharmacokinetic Parameters of Bismuth in Part 2 study.

SECONDARY OUTCOMES:
The percentage of time over a 24-hour period that intragastric pH ≥ 4 and pH ≥ 6 | 1, 14 days
  Percentage of time with intragastric pH ≥ 4 and ≥ 6 during 24-hour monitoring
Proportion of subjects with successful Helicobacter pylori (Hp) eradication | 1, 14 days
  Proportion of subjects with successful Helicobacter pylori (Hp) eradication confirmed by ¹³C-UBT or ¹⁴C-UBT.
Number of subjests With Adverse Events | up to 56 days
  Adverse event severity was graded from 1 to 5 according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Number of subjests With Clinically Notable Electrocardiogram (ECG) Values | up to 56 days
  Record the standard 12-lead ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Lu, Study Director — Shanghai Sinorda Biomedicine Co., Ltd.
Locations (1):
- The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou, China